CLINICAL TRIAL: NCT04112914
Title: Developing an Implementation Strategy for Post-concussion Communication With Low Health Literacy Parents in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Emily Kroshus, Research Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: R21NS111065 (NIH)
Record Dates: First submitted 2019-07-29; First posted 2019-10-02 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Consecutive cohort design with randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education as usual (No Intervention): Participants receive education/healthcare provider communication as usual during their visit to the ED for concussion care.
- New education (Experimental): Participants receive the newly developed educational intervention.
  Interventions: Behavioral: Post-concussion education for families

INTERVENTIONS:
Behavioral: Post-concussion education for families — An educational intervention for families will be developed based on the CDC guidelines for returning to daily activities, school, and sports, adapted with stakeholder feedback to meet the learning needs of low health literacy parents.
  Arms: New education

SUMMARY:
Investigators will conduct a hybrid implementation-effectiveness evaluation of an educational intervention that supports communication with families post-concussion in the emergency department. Primary outcomes will be parent self-report of specific concussion management behaviors two weeks post-visit. Investigators will also explore whether successful implementation is associated with (1) improved parent knowledge and self-efficacy related to helping their child adhere to CDC guidelines for returning to daily activities, school and sports, and (2) decreased disparity in knowledge and self-efficacy between high and low health literacy parents.

DETAILED DESCRIPTION:
Parents can play an important role in evidence-based concussion management by (1) monitoring their child's activity and level of stimulation, (2) communicating with school personnel about potential need for short-term academic accommodations, and (3) ensuring their child does not return to contact or collision sport prematurely and risk greater injury. However, not all parents follow these evidence-based guidelines, in part due to health literacy deficits, and further compounded by the poor fit and inconsistent implementation of educational materials. The initial medical encounter following a concussion provides an important opportunity for evidence-based knowledge translation to parents. Families at risk of low health literacy most often seek initial post-concussion care in emergency departments (ED) and often do not follow-up with a primary care provider or concussion specialist. Knowledge translation to parents in the ED is often inconsistent in terms of content and delivery, and existing approaches often do not meet the needs of families with low health literacy. The Agency for Healthcare Research and Quality's (AHRQ) Re-Engineered Discharge (RED) Toolkit provides an evidence-based approach to supporting the implementation of parent education that has not as yet been adapted for use post-concussion in the ED setting. Investigators will work with stakeholders to develop toolkit to support evidence-based parent education post-concussion in the ED. Guided by the Consolidated Framework for Implementation Research, investigators will adapt the AHRQ RED Toolkit to facilitate post-concussion parent education in the ED. The evidence-based parent education to be shared will be an asynchronous text-based intervention, adapted to meet learning needs of parents with low health literacy and limited English proficiency. Investigators will use parent and provider interviews to iteratively develop the implementation toolkit in consultation with an advisory board comprised of parents. The clinical trial component of the study will be a hybrid implementation-effectiveness evaluation of the educational intervention. Primary outcomes will be parent self-report of specific concussion management behaviors two weeks post-visit. Investigators will also explore whether successful implementation is associated with (1) improved parent knowledge and self-efficacy related to helping their child adhere to CDC guidelines for returning to daily activities, school and sports, and (2) decreased disparity in knowledge and self-efficacy between high and low health literacy parents. Achieving these aims will result in a scalable approach to the implementation of the developed parent education toolkit in the pediatric ED post-concussion. If parents are better able to follow evidence-based guidelines for concussion, they will better advocate and care for their children, and this should improve outcomes for all youth. More broadly, achieving these aims will provide a model for engaging low health literacy parents in adapting evidence-based educational practices for implementation in ED settings.

ELIGIBILITY:
Inclusion criteria:

* Parent/guardian of a child between the ages of 5 and 17 who presented to the Seattle Children's Hospital Emergency Department and was treated for closed head injury.
* Child for whom care was sought was not admitted for inpatient care
* Parent/guardian of child without chronic disease or with non-complex chronic disease
* Parent/guardian with a preferred language for medical care of English or Spanish
* Parent/guardian present in the ED is child's legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital Emergency Department, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were parents in a large pediatric emergency department (ED) whose child (aged 5-17) had sustained a closed head injury in the previous 3 days, was not admitted for inpatient care, and was being discharged. Families waiting for discharge were provided with information about the study. A sequential cohort design (initially control only and then randomization to intervention or control) was used to collect data. The period table presented is for the overall study.
Pre-assignment Details: N/a. All enrolled participants were assigned to the control or intervention condition.
Period: Overall Study
Arm/Group | Education as Usual | New Education
Started | 75 | 23
Completed | 61 | 14
Not Completed | 14 | 9
Not completed — Lost to Follow-up | 13 | 9
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Education as Usual | New Education | Total
Number analyzed (Participants) | 75 | 23 | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.42 (4.98) | 41.36 (4.41) | 40.68 (4.64)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant did not provide sex/gender information.
  Participants
    number analyzed (Participants) | 74 | 23 | 97
    Female | 54 | 16 | 70
    Male | 20 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 2 | 13
  Not Hispanic or Latino | 63 | 21 | 84
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 5 | 0 | 5
  White | 52 | 15 | 67
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 10 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Concussion Management Behaviors: Communication
Description: Parent self-report of specific emotionally supportive concussion management behaviors in the home setting using the emotionally supportive behaviors index. This index is comprised of three communication practices: whether they had talked to their child about "how they are feeling emotionally (e.g., sadness, anxiety)", "the time it takes to recover from a head injury can be different from person to person," and "their concerns about their recovery from head injury." Responses were summed to create a communication index with a possible range of 3 to 9, with higher scores indicating more supportive communication with their child during recovery (Cronbach's alpha=0.59).
Time Frame: Timepoint 3 [Two weeks post-visit]
Population: All participants who responded to concussion management behavior items two weeks post-visit [Cohorts 1 and 2.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Education as Usual | New Education
Number analyzed (Participants) | 61 | 14
Score on a scale | 5.49 (1.68) | 6.71 (2.02)
Statistical Analysis 1: Comparison: Education as Usual vs New Education; Test type: Superiority; p = 0.021, Regression, Linear; Mean Difference (Final Values) = 0.27

2. Primary Outcome: Change in Concussion Management Behaviors: Supportive/Rehabilitation-related
Description: Parent self-report of specific instrumentally-supportive concussion management behaviors in the home setting using the instrumentally supportive behaviors index. This index was comprised of three rehabilitation-related behaviors: "helped child do more physical activity as symptoms improved," "allowed child to return to normal media use as symptoms improved," "and helped child adjust bedtime or sleep environment." Responses were summed to create an instrumental support behavioral index with a possible range of 3 to 9, with higher scores indicating more supportive/rehabilitation-related behaviors (Cronbach's alpha=0.55).
Time Frame: Timepoint 3 [Two weeks post-visit]
Population: All participants who responded to concussion management behavior items two weeks post-visit [Cohorts 1 and 2].
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Education as Usual | New Education
Number analyzed (Participants) | 61 | 14
Score on a scale | 7.35 (1.51) | 7.57 (1.87)
Statistical Analysis 1: Comparison: Education as Usual vs New Education; Test type: Superiority; p = 0.638, Regression, Linear; Mean Difference (Final Values) = 0.06

3. Primary Outcome: Change in Concussion Management Behaviors: Follow-up Appointment
Description: Percentage of participants who reported they had scheduled a follow-up appointment for their child.
Time Frame: Timepoint 3 [Two weeks post-visit]
Population: All participants who responded to concussion management behavior items two weeks post-visit [Cohorts 1 and 2].
Measure: Count of Participants; unit: Participants
Arm/Group | Education as Usual | New Education
Number analyzed (Participants) | 61 | 14
Participants
  Yes | 22 | 7
  No | 39 | 7
Statistical Analysis 1: Comparison: Education as Usual vs New Education; Test type: Superiority; p = 0.338, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [0.55 to 5.72]

4. Secondary Outcome: Change in Concussion Management Self-efficacy: Communication
Description: Self-report of parent confidence in their ability to engage in specific emotionally supportive concussion management behaviors in the home setting using the communication self-efficacy scale. For each of the behaviors, parents were asked to report how challenging it would be to engage in each. Responses were obtained on a 5-point scale where higher scores indicate that performing the behavior would be more challenging (i.e., they have lower self-efficacy). For each domain-specific measure, item level means were calculated, meaning there was a possible range of 1 to 5. In this sample, internal consistency reliability was adequate for the communication subscale (Cronbach's alpha=0.90).
Time Frame: Timepoint 1 [At ED visit], Timepoint 3 [Two weeks post-visit]
Population: All participants who responded to the self-efficacy scale items at Timepoint 1 and Timepoint 3 [Cohort 2 only].
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Education as Usual | New Education
Number analyzed (Participants) | 10 | 14
Score on a scale
  Timepoint 1 | 4.69 (0.57) | 4.71 (0.56)
  Timepoint 3 | 4.80 (0.42) | 4.81 (0.53)
Statistical Analysis 1: Comparison: Education as Usual vs New Education; Test type: Superiority; p = 0.606, Regression, Linear; Mean Difference (Final Values) = 0.13

5. Secondary Outcome: Change in Concussion Management Self-efficacy: Supportive/Rehabilitation-related
Description: Self-report of parent confidence in their ability to engage in specific instrumentally-supportive concussion management behaviors in the home setting using the rehabilitation self-efficacy scale. For each of the parenting behaviors, parents were asked to report how challenging it would be to engage in each. Responses were obtained on a 5-point scale where higher scores indicate that performing the behavior would be more challenging (i.e., they have lower self-efficacy). For each domain-specific measure, item level means were calculated, meaning there was a possible range of 1 to 5. In this sample, internal consistency reliability was adequate for the rehabilitation subscale (Cronbach's alpha=0.79).
Time Frame: Timepoint 1 [At ED visit], Timepoint 3 [Two weeks post-visit]
Population: All participants who responded to the self-efficacy items at Timepoint 1 and Timepoint 3 [Cohort 2 only]
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Education as Usual | New Education
Number analyzed (Participants) | 10 | 14
Score on a scale
  Timepoint 1 | 3.39 (0.55) | 3.48 (0.44)
  Timepoint 3 | 3.28 (0.34) | 3.41 (0.55)
Statistical Analysis 1: Comparison: Education as Usual vs New Education; Test type: Superiority; p = 0.508, Regression, Linear; Mean Difference (Final Values) = 0.12

6. Secondary Outcome: Change in Concussion Management Self-efficacy: Follow-up
Description: Parent self-report of how challenging it would be to make a follow-up appointment for their child. Responses were obtained on a 5-point scale, where higher scores indicate that performing the behavior would be more challenging (i.e., they have lower self-efficacy). Item level means were calculated, meaning there was a possible range of 1 to 5.
Time Frame: Timepoint 1 [At ED visit], Timepoint 3 [Two weeks post-visit]
Population: All participants who responded to the self-efficacy items at Timepoint 1 and Timepoint 3 [Cohort 2 only]
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Education as Usual | New Education
Number analyzed (Participants) | 10 | 14
Score on a scale
  Timepoint 1 | 4.83 (0.53) | 4.77 (0.43)
  Timepoint 3 | 4.70 (0.48) | 5.00 (0.00)
Statistical Analysis 1: Comparison: Education as Usual vs New Education; Test type: Superiority; p = 0.042, Regression, Linear; Mean Difference (Final Values) = 0.45

7. Secondary Outcome: Change in Concussion Knowledge
Description: Self-report of parent knowledge about the benefits of engaging in specific concussion management behaviors in the home setting was measured using the concussion knowledge index. This index was comprised of 10 true or false questions reflecting the knowledge parents need to perform the targeted guideline-consistent communication, rehabilitation, and external engagement behaviors. The index has a potential range of 0-10, with higher scores indicating greater knowledge.
Time Frame: Timepoint 1 [At ED visit], Timepoint 3 [Two weeks post-visit]
Population: All participants who responded to concussion knowledge index items at Timepoint 1 and Timepoint 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Education as Usual | New Education
Number analyzed (Participants) | 61 | 14
Score on a scale
  Timepoint 1 | 6.05 (1.43) | 6.22 (1.68)
  Timepoint 3 | 6.45 (1.68) | 7.29 (1.54)
Statistical Analysis 1: Comparison: Education as Usual vs New Education; Test type: Superiority; p = 0.128, Regression, Linear; Mean Difference (Final Values) = 0.16

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Education as Usual | New Education
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/23
Other Adverse Events (participants affected / at risk) | 0/75 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT04112914/Prot_SAP_000.pdf
  • Informed Consent Form: Cohort 2 (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/14/NCT04112914/ICF_001.pdf
  • Informed Consent Form: Cohort 1 (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT04112914/ICF_002.pdf